CLINICAL TRIAL: NCT03390738
Title: Nivolumab as Treatment for Recurrent/Metastatic Nasopharyngeal Carcinoma After Failing 2 Lines or More Previous Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew funding for Nivolumab
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Dora Kwong, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-1501
Record Dates: First submitted 2017-12-11; First posted 2018-01-04 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravenous nivolumab 240mg (Experimental): Intravenous nivolumab 240mg every 2 weeks until radiologically-documented disease progression, unacceptable toxicity as judged by investigators or patient withdrawal.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Intravenous nivolumab 240mg every 2 weeks until radiologically-documented disease progression, unacceptable toxicity as judged by investigators or patient withdrawal
  Other Names: OPDIVO

SUMMARY:
A phase II, open label, single arm, single agent study using nivolumab in patients who failed 2 or more lines of previous chemotherapy for recurrent/metastatic NPC (At least 1 line should include platinum based chemotherapy)

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic NPC incurable by local therapies and failed at least 2 lines of previous chemotherapy with at least 1 line including platinum based chemotherapy
* Measurable disease (RECIST 1.1)
* ECOG 2 or less
* Life expectancy greater than 3 months
* Adequate organ function
* (Provided tissue for PD-L1 biomarker analysis from a core or excisional biopsy Paired biopsy of baseline tissue at first diagnosis and for recurrence if possible) - optional but encouraged

Exclusion Criteria:

* Suitable for local therapy
* Did not have prior platinum chemotherapy
* Immunodeficiency; immunosuppressive treatment
* Anti-cancer monoclonal antibody treatment within 4 weeks prior to Day 1
* Other cancer treatment within 2 weeks prior to Day 1
* Other malignancies (some exceptions)
* CNS metastases; carcinomatous meningitis
* Active temporal lobe necrosis or on steroid treatment
* Autoimmune disease
* Active, non-infectious pneumonitis
* Active infection requiring systemic treatment
* Hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate of patients. Response will be assessed by RECISTS 1.1 criteria | 1 year

SECONDARY OUTCOMES:
Toxicities as defined by CTCAE criteria | 1 year
  To characterize the safety and tolerability of nivolumab in subjects with recurrent/metastatic NPC. This will be based on subjects who experienced toxicities as defined by CTCAE criteria, receiving at least one dose of nivolumab.

IPD SHARING:
Plan to Share IPD: Undecided